Official Title: A Meditation Intervention on Subconcussive Head Impacts

NCT04225663

IRB-approved date: 7/27/22



You are being asked to sign this addendum because you are participating in a research study at Wake Forest Baptist entitled A Meditation Intervention on Sub-Concussive Head Impacts.

You do not have to sign this addendum to remain in the study.

## **PURPOSE OF THIS ADDENDUM**

The purpose of this addendum is to inform you that your data from the Sway Medical app that obtained your balance and cognitive information will be shared with this study conducted at Wake Forest Baptist.

| Except for the updated information above, the term You will receive a copy of this signed addendum. | s of your original co | nsent form rema | in in full effect |
|---|---|---|---|
| QUESTIONS REGARDING THIS ADDENDUM If you have any questions or concerns regarding this at a contact William Floor If you have any questions, suggestions or concerns | s addendum, please d at). | _ | |
| contact the Institutional Review Board at Forest at | | | |
| STATEMENT OF CONSENT The purpose of this addendum has been explained to questions have been answered to my satisfaction. I below, with the understanding that I may withdraw signed and dated copy of this addendum. | have read this adde | ndum and agree | by signing |
| Subject Name (Printed): | | | |
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent (Printed): | | _ | |
| Person Obtaining Consent: | Date: | Time: | am pm |